CLINICAL TRIAL: NCT00308984
Title: Multi-Center Study on the Incidence of Intra-operative Awareness and Recall in the Pediatric Population Undergoing General Anesthesia: CARE--Childhood Awareness and Recall Evaluation
Brief Title: CARE--Childhood Awareness and Recall Evaluation
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 225
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Anesthesia
Keywords: Pediatrics; Intraoperative Awareness; Pediatric Anesthesia
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the incidence of recall or awareness under anesthesia in children aged 5-15 by collecting anesthetic and post-operative follow-up data relating to intra-operative recall during general anesthesia.

The hypothesis is that the implementation of routine awareness follow-up evaluation in children undergoing general anesthesia will identify that the incidence of intra-operative awareness in children is equal to or greater than in adults.

DETAILED DESCRIPTION:
Awareness, or the unwanted recall of intra-operative events occurring during general anesthesia, is a potentially avoidable anesthetic complication that poses the risk for psychological sequelae. While the reported incidence is 0.1-0.2% in adults, this translates to > 20,000 cases of awareness occurring in adults annually in the United States (Ekman, 2004; Myles, 2000; Sandin, 2000; Sebel, 2004; Myles, 2004). Patients who experience recall may subsequently exhibit post-traumatic stress and psychological symptoms (Sebel, 2004; Myles, 2004; Moerman, 1993; Lennmarken, 2002). Furthermore; studies have shown that up to 54% of adult patients worry about the possibility of awareness during surgery (Klafta, 1996). Subsequent to the recent studies on unintended intraoperative awareness and published data on the impact of Bispectral Index in preventing and detecting anesthesia awareness, the Joint Commission on Accreditation of Healthcare Organizations has classified intraoperative awareness as a sentinel event (2004).

Limited data are available regarding the incidence and consequences of awareness in children. Studies which are available have identified a significantly higher incidence of intraoperative recall in children than has been shown in adults. McKie reported an incidence of 5% factual recall in 202 patients aged 7-14 years in 1973 (1973). The incidence of dreaming was reported as 11%. Hobbs, in 1988, reported a 19% incidence of dreaming and no awareness in 120 pediatric patients who received the "Liverpool anesthetic technique" (N20, O2, relaxant). Ranta reported 0.4% awareness in 4800 patients aged 12 years or older, with the youngest patient demonstrating undisputed awareness at 20 years of age (1998). More recently, Lopez et. al., found an 8% incidence of awareness in children 6-16 years of age, with a significant relationship between multiple attempts to secure the airway and the likelihood of awareness (2004). Most recently, a study published in 2005 by Davidson, et. al., found an incidence of 0.8% in 864 children aged 5-12 years of age with general anesthesia as is practiced in Australia. Likely explanations for more frequent awareness in children include altered anesthetic pharmacology in children and differences in the practice of pediatric anesthesia.

Post-operative behavior changes including emergence delirium, general anxiety, nighttime crying, enuresis, separation anxiety and temper tantrums have been described to occur up in to 50% of children undergoing surgery (Kain, 1996). Studies have also shown a correlation between pre-operative anxiety levels of both the child and parents, and may result in a greater risk of emergence delirium and later maladaptive behaviors. These results have not demonstrated a cause-effect relationship (Kain, 2004). Evaluating for intra-operative awareness or unwanted recall of intra-operative events with or without depth of anesthesia monitoring, may add to the knowledge base for causal factors in postoperative maladaptive behavior changes in the pediatric population.

The JCAHO Sentinel Event Alert, Issue 32, dated October 6, 2004, describes recommendations for health care organizations which perform procedures under general anesthesia, for the prevention and detection of intra-operative awareness. Specific recommendations include: identification of patients who are at higher risk for intraoperative awareness, appropriate follow-up of all patients, including children, who have undergone general anesthesia, and identification, management and, if appropriate, referral of patients who have experienced awareness.

Since little data exists on the incidence and identification of intra-operative awareness in children, this multi-center, prospective, observational, cohort evaluation is being conducted to describe and evaluate the incidence of awareness during routine general anesthetic practice in children. Following IRB approved informed consent (and assent as appropriate), children will sequentially be enrolled to participate in the study. Participating institutions will share de-identified data of enrolled pediatric patients undergoing general anesthesia. Each center will collect and maintain patient data in compliance with all privacy and institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Children 5-15 years of age scheduled for a surgical procedure that requires general anesthesia.
* Children able to respond to and answer post-operative follow-up questions at 3 time intervals post anesthesia: prior to discharge from the post-operative recovery area (or within the first 24 hours following surgery as clinically indicated), 3 (+ 1) days and 14 (+ 2) days post-operatively.
* Ability to speak and understand English.
* Anticipated length of general anesthesia of at least 30 minutes.

Exclusion Criteria:

* Children with known cognitive or neurologic impairment, psychiatric illness or developmental delay consistent with inability to accurately or adequately respond to or answer post-operative follow-up recall questions relating to their anesthesia experience.
* Expectation that the child will remain endotracheally intubated beyond 24 hours postoperatively.
* Anticipated use of ketamine for anesthetic management.
* Children that have had surgery or general anesthesia within the past 6 months or it is anticipated that child will require additional surgeries within the 14 day study follow-up time period.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 5-15 years of age scheduled for a surgical procedure that requires general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 1784 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shobha Malviya, MD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - The Children's Hospital, University of Colorado School of Medicine, Denver, Colorado
  - Children's Hospital of Atlanta at Egleston, Emory University, Atlanta, Georgia
  - Mott Children's Hospital, University of Michigan Health System, Ann Arbor, Michigan

REFERENCES:
- [Background] Ekman A, Lindholm ML, Lennmarken C, Sandin R. Reduction in the incidence of awareness using BIS monitoring. Acta Anaesthesiol Scand. 2004 Jan;48(1):20-6. doi: 10.1111/j.1399-6576.2004.00260.x. PMID 14674969
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Sandin RH, Enlund G, Samuelsson P, Lennmarken C. Awareness during anaesthesia: a prospective case study. Lancet. 2000 Feb 26;355(9205):707-11. doi: 10.1016/S0140-6736(99)11010-9. PMID 10703802
- [Background] Sebel PS, Bowdle TA, Ghoneim MM, Rampil IJ, Padilla RE, Gan TJ, Domino KB. The incidence of awareness during anesthesia: a multicenter United States study. Anesth Analg. 2004 Sep;99(3):833-839. doi: 10.1213/01.ANE.0000130261.90896.6C. PMID 15333419
- [Background] Myles PS, Leslie K, McNeil J, Forbes A, Chan MT. Bispectral index monitoring to prevent awareness during anaesthesia: the B-Aware randomised controlled trial. Lancet. 2004 May 29;363(9423):1757-63. doi: 10.1016/S0140-6736(04)16300-9. PMID 15172773
- [Background] Moerman N, Bonke B, Oosting J. Awareness and recall during general anesthesia. Facts and feelings. Anesthesiology. 1993 Sep;79(3):454-64. doi: 10.1097/00000542-199309000-00007. PMID 8363069
- [Background] Lennmarken C, Bildfors K, Enlund G, Samuelsson P, Sandin R. Victims of awareness. Acta Anaesthesiol Scand. 2002 Mar;46(3):229-31. doi: 10.1034/j.1399-6576.2002.t01-1-460301.x. PMID 11939910
- [Background] Klafta JM, Roizen MF. Current understanding of patients' attitudes toward and preparation for anesthesia: a review. Anesth Analg. 1996 Dec;83(6):1314-21. doi: 10.1097/00000539-199612000-00031. PMID 8942605
- [Background] Preventing, and managing the impact of, anesthesia awareness. Sentinel Event Alert. 2004 Oct 6;(32):1-3. No abstract available. PMID 15470805
- [Background] McKie BD, Thorp EA. Awareness and dreaming during anaesthesia in a paediatric hospital. Anaesth Intensive Care. 1973 Aug;1(5):407-14. doi: 10.1177/0310057X7300100507. No abstract available. PMID 4761535
- [Background] Hobbs AJ, Bush GH, Downham DY. Peri-operative dreaming and awareness in children. Anaesthesia. 1988 Jul;43(7):560-2. doi: 10.1111/j.1365-2044.1988.tb06687.x. PMID 3414918
- [Background] Ranta SO, Laurila R, Saario J, Ali-Melkkila T, Hynynen M. Awareness with recall during general anesthesia: incidence and risk factors. Anesth Analg. 1998 May;86(5):1084-9. doi: 10.1097/00000539-199805000-00035. PMID 9585303
- [Background] Lopez U, Iselin-Chavez I, Habre W. Incidence of awareness during general anaesthesia in children. Br J Anaesth. 2004; 93(3):490P-491P.
- [Background] Davidson AJ, Huang GH, Czarnecki C, Gibson MA, Stewart SA, Jamsen K, Stargatt R. Awareness during anesthesia in children: a prospective cohort study. Anesth Analg. 2005 Mar;100(3):653-661. doi: 10.1213/01.ANE.0000150604.73481.00. PMID 15728046
- [Background] Kain ZN, Caldwell-Andrews AA, Maranets I, McClain B, Gaal D, Mayes LC, Feng R, Zhang H. Preoperative anxiety and emergence delirium and postoperative maladaptive behaviors. Anesth Analg. 2004 Dec;99(6):1648-1654. doi: 10.1213/01.ANE.0000136471.36680.97. PMID 15562048
- [Background] Kain ZN, Mayes LC, O'Connor TZ, Cicchetti DV. Preoperative anxiety in children. Predictors and outcomes. Arch Pediatr Adolesc Med. 1996 Dec;150(12):1238-45. doi: 10.1001/archpedi.1996.02170370016002. PMID 8953995
- [Result] Malviya S, Galinkin JL, Bannister CF, Burke C, Zuk J, Popenhagen M, Brown S, Voepel-Lewis T. The incidence of intraoperative awareness in children: childhood awareness and recall evaluation. Anesth Analg. 2009 Nov;109(5):1421-7. doi: 10.1213/ANE.0b013e3181b620b0. Epub 2009 Aug 27. PMID 19713260